CLINICAL TRIAL: NCT01901718
Title: An Observational, Non-Interventional Trial to Assess Patient Satisfaction and Safety of Subsys™ Spray Compared to Actiq® for the Management of Breakthrough Pain in Chronic Pain Patients.
Brief Title: An Observational, Non-Interventional Trial to Assess Patient Satisfaction and Safety of Subsys™ Spray.
Status: Terminated | Type: Observational
Why Stopped: Enrollment was more challenging than anticipated.
Sponsor: International Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ICRI-Subsys-001
Record Dates: First submitted 2013-04-25; First posted 2013-07-17 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Breakthrough Pain
Keywords: Breakthrough Pain; Subsys; Fentanyl; Opioid; Persistent Pain
MeSH Terms: conditions — Breakthrough Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subsys: Cancer patients experiencing breakthrough pain.

SUMMARY:
Chronic pain patients who experience breakthrough pain in the background of controlled persistent pain with opioids will be followed for 3 months in order to assess the safety and titration trends in the clinical practice setting of a novel fentanyl sublingual spray (Subsys™) for the treatment of breakthrough pain.

DETAILED DESCRIPTION:
Approximately 100 subjects across 10 centers throughout the United States will be enrolled into the study. Subjects who are currently taking Actiq® for their breakthrough pain and will be discontinued due to lack of efficacy, poor tolerability, patient or prescriber dissatisfaction and meet all other study inclusion criteria and none of the exclusion criteria will be candidates to receive a sublingual fentanyl spray (Subsys™). The total duration of the study for each subject will be no more than 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age.
* Subjects who are experiencing 1-4 episodes of break through pain per day in spite of optimized background analgesia and who have taken at least 60 mg/day of morphine (or equivalent analgesic) for at least 7 days.
* Who are currently using Actiq® for their breakthrough pain and are being discontinued due to lack of efficacy, side effects, patient dissatisfaction or prescriber dissatisfaction with treatment.
* Are able to follow and complete all necessary study procedures.
* Are willing and able to give written informed consent before participating in the study.
* Enrolled in the class wide REMS as verified by the study personnel.

Exclusion Criteria:

* Subjects who are not opioid tolerant.
* Using a rapid onset opioid other than Actiq® to manage their breakthrough pain.
* Have physical abnormalities of the floor of the mouth that could affect absorption as determined by investigator.
* Are subjects with uncontrolled or rapidly escalating pain.
* Are subjects with a history of alcohol or substance abuse within the last 3 years.
* Have a clinically significant medical history (past or present) of any disease that would compromise the study or the well-being of the subject.
* Are subjects who have participated in another clinical trial with an analgesic within the last month.
* Are female subjects with a positive pregnancy test or who are currently lactating.
* Are subjects who are taking medications that are known inhibitors of the CYP3A4 isozyme, such as ketoconazole.
* Are subjects who have taken a monoamine inhibitor within 14 days before a dose of study medication.
* Opioid being used for chronic migraine or acute pain.
* Are subjects who are unsuitable for inclusion for any other reason, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain patients who are opioid tolerant and who have failed Actiq® therapy for their breathrough pain will be prescribed Subsys™ fentanyl sublingual spray for their breakthrough pain.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change | 30, 60, 90 days
  The overall impression of change based on a patient's response to the Patient Global Impression of Change (PGIC) questionnaire at month 1, 2, and 3 or upon early discontinuation.

SECONDARY OUTCOMES:
Percent of Patients Satisfied with Treatment | Baseline, 30, 60, 90 days
  Patients will rate their treatment satisfaction using a 5-point scale ranging from 1= Very Dissatisfied to 5= Very Satisfied.
Study Medication Ease of Use | Baseline, 30, 60, 90 days
Quality of Life | Baseline, 30, 60, 90 days
  Short Form 12 Question Health Survey Version 2 (SF-12v2) will be used to assess a subject's general quality of life.
Assessment of Sleep | Baseline, 30, 60, 90 days
  Medical Outcomes Score (MOS) Sleep Subscale will be used to measures 6 dimensions of sleep and is a useful indicator of the efficacy of analgesic medications.
Medication Dosing | Baseline
  Equianalgesic dosing will be calculated based on subject's prior dose of Actiq® and final effective dose of Subsys™.
Weight | Baseline, 30, 60, 90 days
Blood Glucose | Baseline and 90 days
  Blood will be drawn to measure HbA1c.

OTHER OUTCOMES:
Optimal Dose Calculation | 14 Days
  Time to "optimal" dose of an open-label study medication in the Titration phase.

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Nalamachu, MD, Principal Investigator — International Clinical Research Institute
Locations (1):
- International Clinical Research Institute, Overland Park, Kansas, United States